CLINICAL TRIAL: NCT05971771
Title: A Randomized, Double-Blind, Placebo Controlled, Single Center Pilot Study to Assess the Impact of Sleep Supplement on Sleep Health
Brief Title: Study to Assess Impact of Dietary Supplement on Sleep Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmanex (Industry)
Collaborators: Dermatology Consulting Services, High Point NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCS-7-23
Record Dates: First submitted 2023-06-15; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-06

CONDITIONS: Sleep
Keywords: Sleep; Alertness; Restfulness; Dietary AND Supplement
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo controlled, parallel designed study in healthy subjects
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Products will be delivered in forms that it will not be discernable (to participant, investigator, or care provider) as to which product is active or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Sleep Supplement containing Magnesium and Saffron Extract (Experimental): Powder that is to be mixed into 3oz. of water, 30-60 minutes before going to bed
  Interventions: Dietary Supplement: Treatment
- Placebo (Placebo Comparator): Placebo that is 2 softgels that will be taken with water, 30-60 minutes prior to going to bed.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Two softgels to be taken with water that is to be consumed approximately 30-60 minutes before going to bed
  Other Names: Placebo Supplement
  Arms: Placebo
Dietary Supplement: Treatment — 14mg saffron extract and 250mg magnesium citrate that is powder that is mixed in 3-4 oz of water and consumed 30-60 minutes before going to bed
  Other Names: Supplement for supporting sleep
  Arms: Active: Sleep Supplement containing Magnesium and Saffron Extract

SUMMARY:
Sleep is essential for health and wellness. Sleep disruption can occur due to emotional stress, advancing age, hormonal imbalance, medications, and many other causes, some of which are presently unknown. Most pharmaceutical sleep products artificially induce sedation without providing quality sleep. Thus, a need exists for safe dietary supplement to promote and support healthy sleep that will encourage restful sleep. This study will examine the efficacy, tolerance, and safety of sleep supplement as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female 20-60 years of age at the time of informed consent.
* Recorded baseline BMI is ≥18.5 and ≤29.9 kg/m2.
* A score of 5 or higher on the Pittsburgh Sleep Quality Index.
* Willing and able to give informed consent
* Willing to maintain consistent diet and physical activity through the study period.
* Willing to limit alcohol consumption to ≤14 drinks per week, no more than 4 drinks at a time, and no more than 1 drink within 4h of bedtime.
* Willing to limit caffeine consumption to no more than 4 servings per day and no caffeine within 6h of bedtime.

Exclusion Criteria:

* Could not or did not want to participate in clinical study.
* Taken nutritional supplements for sleep or stress in the previous 6 months.
* Have received non-pharmacological treatment for sleep disorders (eg. Cognitive behavioral therapy, relation therapy) in previous 6 months
* Any known allergy or intolerance to any of the ingredients contained in supplement.
* Planned surgical procedure during the course of the study.
* Used nicotine in the past 6 months.
* Have a major psychiatric disorder as determined by the Mini International Neuropsychiatric Inventory
* A history of unconventional sleep pattern, a diagnosed sleep disorder, or chronic medical condition that could affect energy/fatigue levels.
* Consume more than 400mg of caffeine per day in the past 2 weeks.
* Used any psychotropic medications, stimulants, cannabis, non-registered drug products, or illicit substances in the past 4 weeks.
* At risk of drug or alcohol abuse
* Used any sleep aids in the past 2 weeks.
* Employed in night shift work or rotational shift work
* Currently pregnant, nursing, planning to become pregnant, or unwilling to use a medically approved form of contraception will be excluded.
* Individuals who sleep more than 10 hours.
* Typically take a nap during the day.
* Those planning travel or vacation during the study period.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sleep quality index | Baseline, Day 1, Day 7, Day 28
  Change from baseline in validated Pittsburgh Sleep Quality Index (0-21, higher number indicates poorer quality)
Change from baseline sleep duration and quality from diary | Baseline and Daily for 28 days
  Change from baseline with Daily Sleep Diary

SECONDARY OUTCOMES:
Change from baseline perceived stress scale | Baseline, Day 1, Day 7, Day 28
  Change from baseline with validated perceived stress questionnaire
Change from baseline Insomnia severity index | Baseline, Day 1, Day 7, Day 28
  Change from baseline using validated Insomnia Severity Index (0-28, higher number indicates more severe insomnia)
Change from baseline in restorative sleep as measured by Restorative Sleep Questionnaire (RSQ) | Baseline, Day 1, Day 7, Day 28
  Change from baseline using restorative sleep questionnaire as measured by Restorative Sleep Questionnaire (RSQ) that is a 9-item scale/question assessing symptoms over the last week. The total score ranges from 0 to 100, with higher scores indicating better restorative sleep
Change from baseline in mood | Baseline, Day 1, Day 7, Day 28
  Change from baseline using abbreviated Profile of Mood States (POMS) is a widely used questionnaire of 24 items and four scales. Total numbers range from 0-not at all to 4-very strong
Change from baseline in skin attributes | Baseline, Day 7, and Day 28
  Change from baseline in skin attributes using 1-5 scale (1 strongly disagree to 5 strongly agree) with questionnaire regarding skin appearance (youthfulness, glow, evenness, hydration, etc)

OTHER OUTCOMES:
Change in diastolic blood pressure measurement (safety measure) | Baseline and Day 28
  Change from baseline diastolic blood pressure changes using sphygmomanometer
Change in systolic blood pressure measurement (safety measure) | Baseline and Day 28
  Change from baseline systolic blood pressure changes using sphygmomanometer
Change in body weight | Baseline and Day Day 28
  change from baseline in body weight as measured in pounds

IPD SHARING:
Plan to Share IPD: No